CLINICAL TRIAL: NCT04980261
Title: Clinical Trial of Freeze-dried Bovine Hydroxyapatite/Secretome Composite Application for the Management of Long Bone Defects in the Lower Extremities
Brief Title: Freeze-dried Bovine Hydroxyapatite/Secretome Composite for Bone Defects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Soetomo General Hospital (Other Government)
Collaborators: Dr. Ramelan Naval Hospital (Unknown); Airlangga University Hospital (Unknown); Sidoarjo General Hospital (Unknown); Cell & Tissue Bank, Dr. Soetomo General Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0045/KEPK/VIII/2020
Record Dates: First submitted 2021-07-18; First posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-04

CONDITIONS: Bone Loss
Keywords: Bone Defects; Bone Substitutes; Hydroxyapatites; Mesenchymal Stem Cells; Secretome
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Transplantation, Autologous

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (ORIF + autograft) (Active Comparator): The patients will receive the current gold standard to treat long bone defects.
  Interventions: Procedure: ORIF + autograft
- Treatment Group (ORIF + FD BHA/Secretome composite) (Experimental): The patients will receive a novel bone substitute following the ORIF procedure.
  Interventions: Procedure: ORIF + FD BHA/Secretome

INTERVENTIONS:
Procedure: ORIF + autograft — Patients will undergo a standard open reduction internal fixation (ORIF) procedure with autograft implantation (from the iliac crest).
  Arms: Control Group (ORIF + autograft)
Procedure: ORIF + FD BHA/Secretome — Patients will undergo an ORIF procedure and subsequently receive freeze-dried bovine hydroxyapatite/secretome composite implantation.
  Arms: Treatment Group (ORIF + FD BHA/Secretome composite)

SUMMARY:
This clinical trial aims to investigate the efficacy of freeze-dried bovine hydroxyapatite/secretome composite application for the management of long bone defects and other bone healing disorders in the lower extremities.

DETAILED DESCRIPTION:
The gold standard for treating bone defect conditions is autologous bone graft (autograft). Autograft promotes bone healing due to its osteoconductive (serving as a foundation that facilitates bone growth), osteoinductive (stimulates progenitor cells), and osteogenesis (acting as a precursor of osteoblasts and osteoclasts) properties. However, donor site morbidity and persisting pain following harvest remains a major problem. Hence, we attempt to investigate the efficacy of other bone substitutes, i.e., bovine hydroxyapatite/secretome composite, to treat long bone defects and other bone healing disorders in the lower extremities.

Bovine hydroxyapatite (BHA) is a xenograft (animal-derived graft) with osteoconductive properties. Simultaneously, the secretome of the mesenchymal stem cells contains cytokines, chemokines, and growth factors, which possess osteoinductive properties. Thus, we hypothesize that the combination (composite) of BHA/secretome (in the form of freeze-dried (FD) BHA/secretome composite) will promote bone healing ability that is equal to autografts while eliminating donor-site morbidity in the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with bone defects (less than 5 cm) in the diaphysis of the long bones of the lower extremities due to trauma and other bone healing disorders
* No history of comorbid diseases
* Willing to be involved in the clinical trial

Exclusion Criteria:

* Patients with bone defects or impaired bone healing caused by tumors, infections, and metabolic diseases
* Suffered from multiple fractures and multitrauma patients
* Loss to follow-up

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
X-ray evaluation immediately following surgery. | Day-0
  A two-view (anterior-posterior/AP and lateral) radiograph will be taken immediately following surgery. The x-ray evaluation will be carried out by a blinded outcome assessor using a scoring system named Radiographic Union Score (Whelan et al., 2010) to assess bone union based on fracture line, callus, and graft resorption on plain radiograph after fracture. This score ranges from 4 to 12, with a higher score indicating a more favorable outcome (better bone healing).
X-ray evaluation at 4 weeks following surgery | 4 weeks
  A two-view (anterior-posterior/AP and lateral) radiograph will be taken immediately following surgery. The x-ray evaluation will be carried out by a blinded outcome assessor using a scoring system named Radiographic Union Score (Whelan et al., 2010) to assess bone union based on fracture line, callus, and graft resorption on plain radiograph after fracture. This score ranges from 4 to 12, with a higher score indicating a more favorable outcome (better bone healing).
X-ray evaluation at 8 weeks following surgery. | 8 weeks
  A two-view (anterior-posterior/AP and lateral) radiograph will be taken immediately following surgery. The x-ray evaluation will be carried out by a blinded outcome assessor using a scoring system named Radiographic Union Score (Whelan et al., 2010) to assess bone union based on fracture line, callus, and graft resorption on plain radiograph after fracture. This score ranges from 4 to 12, with a higher score indicating a more favorable outcome (better bone healing).
X-ray evaluation at 12 weeks following surgery. | 12 weeks
  A two-view (anterior-posterior/AP and lateral) radiograph will be taken immediately following surgery. The x-ray evaluation will be carried out by a blinded outcome assessor using a scoring system named Radiographic Union Score (Whelan et al., 2010) to assess bone union based on fracture line, callus, and graft resorption on plain radiograph after fracture. This score ranges from 4 to 12, with a higher score indicating a more favorable outcome (better bone healing).
X-ray evaluation at 16 weeks following surgery. | 16 weeks
  A two-view (anterior-posterior/AP and lateral) radiograph will be taken immediately following surgery. The x-ray evaluation will be carried out by a blinded outcome assessor using a scoring system named Radiographic Union Score (Whelan et al., 2010) to assess bone union based on fracture line, callus, and graft resorption on plain radiograph after fracture. This score ranges from 4 to 12, with a higher score indicating a more favorable outcome (better bone healing).
Ultrasonography evaluation at 2 weeks | 2 weeks
  A blinded outcome assessor will perform ultrasonography (USG) evaluation to assess the four stages of the bone healing process using a scoring system named Sonographic Union Score developed by our institution. We will evaluate the following parameters: (1) hematoma organization, (2) neovascularization, (3) bone fracture tip echogenicity, (4) bone fracture border, (5) bridging callus echogenicity, (6) bone to bone graft junction gap, (7) callus formation mineralization, (8) bone surface continuity.
Ultrasonography evaluation at 4 weeks | 4 weeks
  A blinded outcome assessor will perform ultrasonography (USG) evaluation to assess the four stages of the bone healing process using a scoring system named Sonographic Union Score developed by our institution. We will evaluate the following parameters: (1) hematoma organization, (2) neovascularization, (3) bone fracture tip echogenicity, (4) bone fracture border, (5) bridging callus echogenicity, (6) bone to bone graft junction gap, (7) callus formation mineralization, (8) bone surface continuity.
Ultrasonography evaluation at 8 weeks | 8 weeks
  A blinded outcome assessor will perform ultrasonography (USG) evaluation to assess the four stages of the bone healing process using a scoring system named Sonographic Union Score developed by our institution. We will evaluate the following parameters: (1) hematoma organization, (2) neovascularization, (3) bone fracture tip echogenicity, (4) bone fracture border, (5) bridging callus echogenicity, (6) bone to bone graft junction gap, (7) callus formation mineralization, (8) bone surface continuity.
Ultrasonography evaluation at 12 weeks | 12 weeks
  A blinded outcome assessor will perform ultrasonography (USG) evaluation to assess the four stages of the bone healing process using a scoring system named Sonographic Union Score developed by our institution. We will evaluate the following parameters: (1) hematoma organization, (2) neovascularization, (3) bone fracture tip echogenicity, (4) bone fracture border, (5) bridging callus echogenicity, (6) bone to bone graft junction gap, (7) callus formation mineralization, (8) bone surface continuity.
Ultrasonography evaluation at 16 weeks | 16 weeks
  A blinded outcome assessor will perform ultrasonography (USG) evaluation to assess the four stages of the bone healing process using a scoring system named Sonographic Union Score developed by our institution. We will evaluate the following parameters: (1) hematoma organization, (2) neovascularization, (3) bone fracture tip echogenicity, (4) bone fracture border, (5) bridging callus echogenicity, (6) bone to bone graft junction gap, (7) callus formation mineralization, (8) bone surface continuity.

SECONDARY OUTCOMES:
Functional evaluation at 8 weeks following surgery. | 8 weeks
  The functional evaluation will be assessed by using a scoring system named LEFS (Lower Extremity Functional Scale). LEFS is a widely known and validated patient-reported outcome measures (PROM) comprising 20 questions that is used to assess lower extremity functions. The patients will be asked to rate the activity listed from 0 to 4 (0 refers to an extreme difficulty/unable to perform activity, while 4 refers to having no difficulty at all). A higher score (maximum 80 points) indicates a very high function (i.e., a more favorable outcome).
Functional evaluation at 12 weeks following surgery. | 12 weeks
  The functional evaluation will be assessed by using a scoring system named LEFS (Lower Extremity Functional Scale). LEFS is a widely known and validated patient-reported outcome measures (PROM) comprising 20 questions that is used to assess lower extremity functions. The patients will be asked to rate the activity listed from 0 to 4 (0 refers to an extreme difficulty/unable to perform activity, while 4 refers to having no difficulty at all). A higher score (maximum 80 points) indicates a very high function (i.e., a more favorable outcome).
Functional evaluation at 16 weeks following surgery. | 16 weeks
  The functional evaluation will be assessed by using a scoring system named LEFS (Lower Extremity Functional Scale). LEFS is a widely known and validated patient-reported outcome measures (PROM) comprising 20 questions that is used to assess lower extremity functions. The patients will be asked to rate the activity listed from 0 to 4 (0 refers to an extreme difficulty/unable to perform activity, while 4 refers to having no difficulty at all). A higher score (maximum 80 points) indicates a very high function (i.e., a more favorable outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Soetomo General Hospital, Surabaya, East Java, Indonesia